CLINICAL TRIAL: NCT01885455
Title: Improving Resection Rates Among African Americans With NSCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00031268; REBAWF 01414 (Other: NCI)
Record Dates: First submitted 2013-06-17; First posted 2013-06-25 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Arm (Active Comparator): Participants who are assigned to the usual care arm may receive the following services: complete staging work-up (CT/PET scan and possible mediastinoscopy), surgical consultation with a general or cardiothoracic surgeon, cardiac clearance and/or pulmonary function testing (if deemed necessary by the evaluating surgeon), surgical resection (wedge resection, lobectomy, pneumonectomy, or radiosurgery, as indicated by the size and location of the tumor), and adjuvant therapy (radiotherapy and/or chemotherapy, as determined by the intraoperative findings and pathology results).
  Interventions: Other: Usual Care
- Intervention Arm (Experimental): The PN will provide each patient with a copy of the NCI's "What You Need to Know About Lung Cancer" booklet and encourage them to re-contact his/her primary care physician (or the physician who diagnosed their probable/proven NSCLC) to discuss treatment options.
  The PNs will provide patients with their contact information and brief patients on their role. The PNs will navigate study participants for up to 4 months (16 weeks, 112 days) after NSCLC diagnosis, until the patient is deemed ineligible for LDTCI (i.e., lung resection or SBRT) by their physician(s), until receipt of LDTCI, or death (whichever comes first).
  During the EPDPN intervention period, PNs will contact each intervention group participant by telephone (or in-person) on weekly basis (at minimum).
  Interventions: Other: Intervention Arm

INTERVENTIONS:
Other: Usual Care — Usual care includes: complete staging work-up (CT/PET scan and possible mediastinoscopy), surgical consultation with a general or cardiothoracic surgeon, cardiac clearance and/or pulmonary function testing (if deemed necessary by the evaluating surgeon), surgical resection (wedge resection, lobectomy, pneumonectomy, or radiosurgery, as indicated by the size and location of the tumor), and adjuvant therapy (radiotherapy and/or chemotherapy, as determined by the intraoperative findings and pathology results).
  Arms: Usual Care Arm
Other: Intervention Arm — The proposed Intervention (EPDPN) will be administered by the PNs at the intervention sites on an outpatient basis. Several defining, fundamental characteristics of the PNs will ensure consistency of the intervention delivery across the various study sites.
  Arms: Intervention Arm

SUMMARY:
This is a randomized, interventional trial in which the navigation is the intervention. Phase is not applicable. The study is a randomized trial to evaluate the impact of a nurse-led patient navigation intervention in improving rates of receipt of lung-directed therapy with curative intent (LDTCI) among African Americans with early stage lung cancer. Study sites are cluster-randomized to either the usual care study arm or the to the navigation intervention study arm. Randomization occurred at the level of the study site rather than at the level of individual participants. There are two arms.

DETAILED DESCRIPTION:
The burden to participants will be minimized to enhance retention. Patients in the usual care arm receive the current "gold standard" of treatment. The patients in the intervention arm are assigned to a PN, who helps to reduce the barriers to care that could negatively impact the patients' receipt of LDTCI. The telephone-administered survey is administered to all study participants at baseline and at 3-, 6-, and 12-months post-enrollment. It takes approximately 30-40 minutes to administer. The telephone mode of survey administration was chosen to reduce the number of visits that would be required by each patient. Interviews are scheduled at the convenience of the study participants. To further reduce burden to the study participants, the interviewers offer breaks during the interview process. Patients in both arms undergo standard therapy visits. Patients in the navigation arm receive standard therapy visits plus the navigation intervention. Outside of the standard therapy visits, no additional clinic visits are required of the study participants.

Once informed consent has been obtained and the informed consent document is received, the SSC/PN will communicate to the MUSC HCC study staff the participant's contact information and that the participant is ready for baseline survey administration. All the study surveys will be administered by trained MUSC HCC study staff via telephone. A survey answer guide will be provided to the participant either in-person or via mail prior to administration of the baseline survey.

ELIGIBILITY:
Inclusion Criteria:

* AA race
* Clinically suspicious or biopsy-proven, early stage NSCLC, and
* Ages 21 years and older

Exclusion Criteria:

* Previous history of lung cancer
* Spread of newly diagnosed probably/proven lung cancer to other part of the body
* Diagnosis of synchronous cancer other than non-melanoma skin cancer or lung cancer, and
* Receipt of surgical resection or radiosurgery for lung cancer since diagnosis with probable/proven lung cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Receipt of LDTCI | 12 Months Post-Enrollment
  Receipt of lung-directed therapy with curative intent (LDTCI), Inquiry at time of follow-up survey, confirmed by medical record review

SECONDARY OUTCOMES:
Receipt of Surgical and/or Radiation Oncology Consultation Confirmed by Medical Record Review | Baseline, 3, 6, 9, and 12 Months Post-Enrollment
  • Receipt of surgical and/or radiation oncology consultation (defined as outpatient or inpatient consultation with a general or cardiothoracic surgeon and/or radiation oncologist to discuss LDTCI for NSCLC within 4 months post-diagnosis of probable/proven, early stage NSCLC).
Time to LDTCI (For Pts. Who Received LDTCI Only) Confirmed by Medical Record Review | Baseline, 3, 6, 9, and 12 Months Post-Enrollment
  Time to LDTCI (For Pts. Who Received LDTCI Only). Inquiry at Time of Follow-Up Survey, Confirmed by Medical Record Review. Baseline, 3, 6, 9, and 12 Months Post-Enrollment
Satisfaction with Care Received, Patient Satisfaction(REF) (28 items) | 6 Months Post-Enrollment
  Satisfaction with Care Received, Patient Satisfaction(REF) (28 items). 6 Months Post-Enrollment
Time of Death, Follow-up Survey, Confirmed by Medical Record Review | Baseline, 3, 6, 9, and 12 Months Post-Enrollment
  Time of Death. Inquiry at Time of Follow-Up Survey, Confirmed by Medical Record Review , inquiry of cancer registries at study sites, and inquiry of Social Security Death Index. Baseline, 3, 6, 9, and 12 Months Post-Enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Weaver, PhD, Principal Investigator — Wake Forest Universith Health Sciences
Locations (10):
- United States (10):
  - Beebe Healthcare Tunnell Cancer Center, Lewes, Delaware
  - Saint Joseph's/Candler Hospital, Savannah, Georgia
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Ochsner NCORP, New Orleans, Louisiana
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Metro-Minnesota NCORP, Saint Louis Park, Minnesota
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Fox Chase, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT01885455/ICF_000.pdf